CLINICAL TRIAL: NCT05016609
Title: Same-visit Hepatitis C Testing and Treatment to Accelerate Cure Among People Who Inject Drugs: a Cluster Randomised Control Trial (The QuickStart Study)
Brief Title: Same-visit Hepatitis C Testing and Treatment (The QuickStart Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HREC/64731/Alfred-2020-217547
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; velpatasvir

STUDY DESIGN:
Intervention Model Description: A cluster cross-over randomised controlled trial with cluster randomisation performed at the site level. Each site will be randomised to one of the three interventions and one standard of care period. All participants will receive the intervention or comparator that has been allocated to the service they present at.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- POC HCV antibody group (Arm A) (Experimental): This group will receive POC HCV antibody testing via fingerprick using the OraQuick HCV antibody test (OraSure) in addition to the standard-of-care whole-blood conventional laboratory-based HCV PCR viral load testing. Follow up and management of any treatment will be through usual standard-of-care. Participants in this group will also fill out a short behavioural questionnaire and a clinical questionnaire.
  Interventions: Device: OraQuick HCV Antibody test (OraSure Technologies, Inc)
- POC HCV RNA group (Arm B) (Experimental): This group will receive POC HCV antibody testing using the OraQuick HCV antibody test. Participants in this group who return a positive POC HCV antibody result will receive POC HCV viral load testing via fingerstick using the Xpert HCV Viral Load Finger-stick Point-of-Care test (Cepheid) in addition to the standard-of-care whole-blood conventional laboratory-based HCV PCR viral load testing. Follow up and management of any treatment will be through usual standard-of-care. Participants in this group will also fill out a short behavioural questionnaire and a clinical questionnaire.
  Interventions: Device: OraQuick HCV Antibody test (OraSure Technologies, Inc); Device: Xpert HCV Viral Load Finger-stick Point-of-Care test (Cepheid)
- Test and treat group (ArmC) (Experimental): This group will receive POC HCV antibody testing using the OraQuick HCV antibody test. Participants in this group who return a positive POC HCV antibody result will be provided a starter pack of HCV treatment (epclusa). POC tests results will be confirmed through standard-of-care whole-blood conventional laboratory-based HCV PCR viral load testing. HCV RNA positive participants will continue treatment. Participants in this group will also fill out a short behavioural questionnaire and a clinical questionnaire.
  Interventions: Device: OraQuick HCV Antibody test (OraSure Technologies, Inc); Drug: Sofosbuvir/Velpatasvir (Gilead)
- Control (No Intervention): This group will receive the standard of care for HCV testing and treatment. Participants in this group will fill out a short behavioural questionnaire and a clinical questionnaire.

INTERVENTIONS:
Device: OraQuick HCV Antibody test (OraSure Technologies, Inc) — The OraQuick HCV test is a point of care antibody test for detecting HCV antibodies in fingerstick blood. The test takes 20 minutes to provide a result. Appropriate pre- and post-test counselling will be provided to participants.
  Arms: POC HCV RNA group (Arm B); POC HCV antibody group (Arm A); Test and treat group (ArmC)
Device: Xpert HCV Viral Load Finger-stick Point-of-Care test (Cepheid) — Xpert® HCV VL Fingerstick is an in vitro reverse transcription polymerase chain reaction (RT-PCR) assay for the detection and quantification of Hepatitis C Virus (HCV) RNA in human venous and capillary fingerstick EDTA whole blood. Only participants who return a reactive OraQuick HCV Antibody test will be offered the Xpert® HCV VL Fingerstick test. Appropriate pre- and post-test counselling will be provided to participants.
  Arms: POC HCV RNA group (Arm B)
Drug: Sofosbuvir/Velpatasvir (Gilead) — Participants with a detectable HCV antibody will be offered treatment with sofosbuvir/velpatasvir.
  Arms: Test and treat group (ArmC)

SUMMARY:
The QuickStart study aims to assess the impact of three models of HCV care on HCV treatment uptake and cure among people who inject drugs. Rapid point-of-care (POC) HCV testing and test-and-treat strategies will be utilised in primary health care settings across Australia.

DETAILED DESCRIPTION:
The QuickStart Study will explore models of point-of-care HCV testing and a same-day test and treat model to determine the impact of these models on HCV treatment initiation and cure. The study is a cluster cross-over randomised controlled trial. Sites are primary care services in Australia who provide services to people who inject drugs (PWID) and who routinely prescribe treatment for hepatitis C. Clinical services with a primary care practitioner and/or nurse experienced in providing DAA treatment to high numbers of PWID will be recruited to the study. A total of 30 services will be recruited with each service enrolling approximately 60 participants across an intervention and control period. Key participant eligibility include a history of injecting drug use and no previous treatment for HCV with direct acting antivirals.

Each site will participate in a control comparison period in addition to one of three interventions. The three interventions involve:

A) A rapid HCV antibody test using a fingerprick sample and for anybody subsequently diagnosed with hepatitis C, management and treatment will be according to standard of care.

B) A rapid HCV antibody test followed by a POC HCV RNA test for those who return a reactive antibody result. Both these will use a fingerprick sample and for anybody diagnosed with hepatitis C, management and treatment will be according to standard of care.

C) A rapid HCV antibody test using a fingerprick sample and for participants who return a reactive result, an initial starter pack of DAA prior to a confirmed HCV RNA diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* current or former PWID (i.e., injected drugs at least once)
* aged 18 years or over
* attending a participating PHC for any reason
* no previous treatment with DAAs for HCV
* failed interferon based treatment for HCV in the past (i.e., did not achieve cure)
* Medicare eligible
* able to speak and understand English

Exclusion Criteria:

* women known to be currently pregnant or who are breastfeeding
* individuals self-reporting to be currently engaged in treatment for HCV
* unable to provide informed consent
* tested for HCV in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
HCV treatment | Within 12 weeks of enrolment
  The number of participants who start HCV treatment in each of the intervention arms (Arm A, Arm B or Arm C) within 12 weeks of enrolment, compared with standard care testing and treatment (Control Arm).
HCV cure | HCV cure will be measured between 4 and 20 weeks post treatment completion.
  The number of participants who achieve HCV cure in each of the intervention arms (Arm A, Arm B or Arm C), compared with standard care testing and treatment (Control Arm).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Doyle, MBBS, PhD, Principal Investigator — Burnet Institute
Locations (6):
- Australia (6):
  - Mediclinic Australia, Clayton South, Victoria
  - Innerspace, Collingwood, Victoria
  - Corio Community Health Centre, Corio, Victoria
  - Cohealth Fitzroy, Fitzroy, Victoria
  - Homeless Healthcare, Highgate, Western Australia
  - Cockburn Wellbeing, Success, Western Australia

IPD SHARING:
Plan to Share IPD: No
Requests for data sharing can be made to the principal investigator; further approval by the Human Research Ethics Committee may be necessary given the sensitive behaviour and risk information collected in the context of a trial of people who use drugs and hepatitis C testing.

REFERENCES:
- [Derived] Heath K, Guzman R, Elsum I, Wade AJ, Allardice K, Kasza J, Bryant M, Thompson AJ, Stoove M, Snelling T, Scott N, Spelman T, Anderson DA, Richmond J, Howell J, Andric N, Dietze P, Higgs P, Sacks-Davis R, Forbes A, Hellard ME, Pedrana AE, Doyle JS. Balancing Efficiency and Accuracy in Hepatitis C Rapid Antibody Testing: Insights From a Cluster Randomised Crossover Trial. J Viral Hepat. 2025 Aug;32(8):e70043. doi: 10.1111/jvh.70043. PMID 40607684
- [Derived] Doyle JS, Heath K, Elsum I, Douglass C, Wade A, Kasza J, Allardice K, Von Bibra S, Chan K, Camesella B, Guzman R, Bryant M, Thompson AJ, Stoove MA, Snelling TL, Scott N, Spelman T, Anderson D, Richmond J, Howell J, Andric N, Dietze PM, Higgs P, Sacks-Davis R, Forbes AB, Hellard ME, Pedrana AE. Same-visit hepatitis C testing and treatment to accelerate cure among people who inject drugs (the QuickStart Study): a cluster randomised cross-over trial protocol. BMJ Open. 2024 Jul 2;14(7):e083502. doi: 10.1136/bmjopen-2023-083502. PMID 38960465